CLINICAL TRIAL: NCT06148077
Title: Effects of Manual Therapy on Oral Opening, Swallow Function, and Upper Quarter Mobility in Chilean Survivors of Head and Neck Cancer: A Study Protocol for a Controlled, Randomized Study (MATEO Study, MAnual ThErapy for Oral Opening).
Brief Title: Manual Therapy on Oral Opening, Swallow Function and Upper Quarter Mobility on Head and Neck Cancer Survivors
Acronym: MaTeO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Barbara Burgos Mansilla, PhD, Universidad de La Frontera
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DIM23-0023
Record Dates: First submitted 2023-11-17; First posted 2023-11-28 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Cancer; Trismus; Dysfunction
MeSH Terms: conditions — Head and Neck Neoplasms; Trismus | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual Therapy (Experimental): Manual Therapy-based intervention: the session will be performed with the patient in a supine position. If they cannot reach this position, it can be done with the patient sitting in a chair to receive the treatment. The selected maneuvers will focus on cervical, masticatory, and shoulder regions. Besides, intraoral maneuvers will be made using latex gloves, for masseter, medial, and lateral pterygoid muscles. Subsequently, motor control exercises will be performed
  Interventions: Other: Manual Therapy
- Motor Control (Active Comparator): Motor control (exercise): the session will focus on strengthening and stretching exercises for the cervical, masticatory, and shoulder muscles .
  Interventions: Other: Motor control exercises

INTERVENTIONS:
Other: Manual Therapy — 3 times a week, for 6 weeks.
  Arms: Manual Therapy
Other: Motor control exercises — 3 times a week, for 6 weeks.
  Arms: Motor Control

SUMMARY:
Trismus has been reported as the second most common comorbidity in survivors of head and neck cancer (HNC). It is mainly associated with post-radiotherapy subcutaneous fibrosis, muscular atrophy, damage to neurological structures in the neck, or a combination of all, affecting masticatory musculature. In addition to this, the loss of flexibility and strength in the shoulder has also been shown to be related to deficits in the function and quality of life of these patients.

The goal of this clinical trial is to determinate the effectiveness and safety of Manual Therapy (MT) on Oral Opening, Swallow Function, as well as the mobility of the upper quarter, the strength of cervical musculature, pain, functionality, and the perception of quality of life in head and neck cancer survivors.

Participants will be assigned randomly to the study groups: a) manual therapy program and control motor exercises and b) motor control exercises (usual care).

The assessment refers to a baseline form (at the beginning of the study), at 6 weeks and at 6 weeks of patient follow-up.

DETAILED DESCRIPTION:
Manual therapy program consists of 3 sessions a week during 6 weeks, with a total of 18 appointments. Measurements are done before starting, after the last intervention and 6 weeks after finishing the treatment.

ELIGIBILITY:
Inclusion Criteria:

* individuals with HNC
* individuals over 18 years of age
* individuals who have undergone oncological surgery of the head and neck and/or radiotherapy
* having finished oncological medical treatment between 3 and 36 months before inclusion
* having a medical diagnosis of trismus and/or TMD and/or cervical or shoulder dysfunction
* Spanish native speakers

Exclusion Criteria:

* sequelae of previous stroke
* structural instability and/or osteoporosis of the cervical spine, spondylosis, cervical herniated discs
* active osteoradionecrosis or open wounds (fistulas, soft tissue necrosis) in the anatomical treatment area
* tracheostomized individuals
* metastasis or active cancer
* refuse to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Maximal mouth opening (MMO) | 6 weeks
  MMO will be assessed with a sliding calliper measuring the inter-incisor distance asking the patients to open the mouth as maximum as possible.
Temporomandibular disorders (TMD) | 6 weeks
  TMD will be assessed with the Fonseca Anamneses Index, that classifies TMD as no dysfunction, light dysfunction, moderate dysfunction or severe dysfunction
Swallowing function | 6 weeks
  Eating Assessment Tool (EAT-10) will be used to evaluate self-reported swallowing impairments. It is a 5 point Likert scale rating from no impairment to severe problem. The sum of all items contained on the questionnaire is used as the overall score, suggesting an abnormal swallowing when score is higher than 3
Swallowing difficulty | 6 weeks
  A Visual Analogue Scale (VAS) will be used to register swallowing difficulties, ranging from 0 (no problems) to 10 (impossible to swallow)
Dysphagia | 6 weeks
  Water Swallow Test, subject will be ask to drink 100 mL of water as quickly as is comfortably possible. The time to swallow this 100 mL (in seconds) and the number of swallows will be count.

SECONDARY OUTCOMES:
Shoulder active range of motion (AROM) | 6 weeks
  The active range of motion (AROM) of flexion, abduction, and external and internal rotations will be assessed bilaterally. For measurement, a manual goniometer with two arms and a range of 360º will be used.
Cervical active range of motion (AROM) | 6 weeks
  The active range of motion (AROM) of cervical flexion, extension, lateral flexion, and rotation will be assessed. For this purpose, a cervical range of motion instrument (CROM) will be used.
Deep cervical flexors endurance | 6 weeks
  Endurance of deep cervical flexor muscles will be assessed with the deep cervical flexor endurance test, with the patient in a supine lying position with the examiner's hands under his/her head and being told to fold the chin completely to the sternum and raising the head as minimum as possible without touching examiner's hands. Time is counted from when the patient lift his/her head until when he/she can no longer maintain the position.
Muscle Function Test | 6 weeks
  Defined for the upper fibers of the trapezius, will be used as a test to assess shoulder muscle strength. With the subject in a seated position and arms at both sides of the trunk, they will be asked to push caudally-cranially against the evaluator's hand, placed on their shoulder. The muscle function scale ranges from 0 (complete absence of muscle contraction) to 5 (normal muscle response)
Isometric handgrip strength | 6 weeks
  A digital dynamometer with adjustable grip will be used to assess handgrip strength. The patient will be asked, while in a seated position, holding a dynamometer, with the elbow flexed at 90° and the shoulder in a neutral position, to perform a grip with maximum effort. Three attempts will be made with each hand (a total of 6 attempts), with a 1-minute rest between each attempt. The average of the three attempts will be calculated for data analysis.
Pain Intensity | 6 weeks
  At the cervical and temporomandibular joint levels (bilaterally), assessment will be conducted using a validated Visual Analog Scale (VAS): a horizontal line measuring 10 cm in length, with "no pain" at its left end (score 0) and "maximum pain" at its right end (score 10). Patients will be asked to mark the intensity of perceived pain during their day-to-day activities by placing a cross on the line.
Pressure pain thresholds | 6 weeks
  Pressure algometry will be assessed over the temporalis, masseter, upper trapezius and levator scapulae muscles and the C5-C6 zygapophyseal joint, the sternoclavicular joint and the tibialis anterior muscle as a distant reference muscle.Each point to be evaluated will be analyzed three times with a 30-second interval between assessments, and the arithmetic mean of the three measurements will be used for subsequent statistical analysis.
Shoulder pain and disability perception | 6 weeks
  Shoulder pain and disability index (SPADI) will be used to evaluate pain and disability perception of the patients at shoulder level.
Health-related quality of life | 6 weeks
  Questionnaire EORTC QLQ-C30 will be used for measuring quality of life
Health-related quality of life 2 | 6 weeks
  Questionnaire EORTC QLQ-H&N43 will be used for measuring quality of life specifically in survivors of head and neck cancer
Physical Fitness | 6 weeks
  International Fitness Scale (IFIS) will be used to evaluate perceived physical fitness. It contains 4 physical fitness elements (cardiorespiratory endurance, muscular strength, speed/agility and flexibility) to categorize into 5 options, from very poor to very good
Satisfaction with the treatment | 6 weeks
  It will be determined through a pre-designed questionnaire consisting of 6 items, including 1 item for overall satisfaction with scores ranging from 0 to 10, and 5 dichotomous response items (yes/no), where the patient can provide reasons for their response. This instrument has been previously used for this purpose.
Adverse Events (AE) | 6 weeks
  Safety will be recorded in terms of adverse events, defined as any unfavorable change in health that occurs during the intervention. Each adverse event will be characterized based on severity (Grade 1 [mild] to 5 [death]), expectation (expected or unexpected), and potential relationship with study participation (unrelated, possibly related, or related to the study) using the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Burgos, PhD, Principal Investigator — Universidad de La Frontera
Locations (2):
- Chile (2):
  - Barbara Burgos Mansilla, Temuco, Cautin
  - Universidad de La Frontera, Temuco, Cautin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wissinger E, Griebsch I, Lungershausen J, Foster T, Pashos CL. The economic burden of head and neck cancer: a systematic literature review. Pharmacoeconomics. 2014 Sep;32(9):865-82. doi: 10.1007/s40273-014-0169-3. PMID 24842794
- [Background] Parke SC, Langelier DM, Cheng JT, Kline-Quiroz C, Stubblefield MD. State of Rehabilitation Research in the Head and Neck Cancer Population: Functional Impact vs. Impairment-Focused Outcomes. Curr Oncol Rep. 2022 Apr;24(4):517-532. doi: 10.1007/s11912-022-01227-x. Epub 2022 Feb 19. PMID 35182293
- [Background] Kamstra JI, Jager-Wittenaar H, Dijkstra PU, Huisman PM, van Oort RP, van der Laan BF, Roodenburg JL. Oral symptoms and functional outcome related to oral and oropharyngeal cancer. Support Care Cancer. 2011 Sep;19(9):1327-33. doi: 10.1007/s00520-010-0952-4. Epub 2010 Aug 13. PMID 20706851
- [Background] McMillan H, Barbon CEA, Cardoso R, Sedory A, Buoy S, Porsche C, Savage K, Mayo L, Hutcheson KA. Manual Therapy for Patients With Radiation-Associated Trismus After Head and Neck Cancer. JAMA Otolaryngol Head Neck Surg. 2022 May 1;148(5):418-425. doi: 10.1001/jamaoto.2022.0082. PMID 35297966
- [Background] Ortiz-Comino L, Martin-Martin L, Galiano-Castillo N, Castro-Martin E, Fernandez-Gualda MA, Lozano-Lozano M, Fernandez-Lao C. The effects of myofascial induction therapy in survivors of head and neck cancer: a randomized, controlled clinical trial. Support Care Cancer. 2022 Dec 17;31(1):49. doi: 10.1007/s00520-022-07482-9. PMID 36526871
- [Background] Castro-Martin E, Galiano-Castillo N, Fernandez-Lao C, Ortiz-Comino L, Postigo-Martin P, Arroyo-Morales M. Myofascial Induction Therapy Improves the Sequelae of Medical Treatment in Head and Neck Cancer Survivors: A Single-Blind, Placebo-Controlled, Randomized Cross-Over Study. J Clin Med. 2021 Oct 27;10(21):5003. doi: 10.3390/jcm10215003. PMID 34768520
- [Background] Pauli N, Fagerberg-Mohlin B, Andrell P, Finizia C. Exercise intervention for the treatment of trismus in head and neck cancer. Acta Oncol. 2014 Apr;53(4):502-9. doi: 10.3109/0284186X.2013.837583. Epub 2013 Oct 31. PMID 24175896
- [Background] Pattanshetty RB, Patil SN. Role of Manual Therapy for Neck Pain and Quality of Life in Head and Neck Cancer Survivors: A Systematic Review. Indian J Palliat Care. 2022 Jan-Mar;28(1):99-112. doi: 10.25259/IJPC_10_2021. Epub 2021 Dec 18. PMID 35673382
- [Derived] Burgos-Mansilla B, Schneeberger-Hitschfeld P, Astete-Barra K, Mendez-Rojas A, Ortiz-Comino L. Effects of manual therapy on oral opening, swallow function and upper quarter mobility in Chilean survivors of head and neck cancer: a study protocol for a controlled, randomised study (MAnual ThErapy for Oral Opening (MATEO) study). BMJ Open. 2025 Sep 2;15(9):e097131. doi: 10.1136/bmjopen-2024-097131. PMID 40897487